CLINICAL TRIAL: NCT06803745
Title: A Randomized Phase II Trial of Standard-of-Care Reduced-Intensity Conditioning (RIC) With 200 Versus 400 cGy of Total Body Irradiation (TBI) in Patients With Acute Leukemia Undergoing First Allogeneic Blood or Marrow Transplantation (BMT)
Brief Title: Standard-of-Care Reduced-Intensity Conditioning (RIC) With 200 Versus 400 cGy of Total Body Irradiation (TBI) in Patients With Acute Leukemia Undergoing First Allogeneic Blood or Marrow Transplantation (BMT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J24142; IRB00479809 (Other: JHU IRB)
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Acute Leukemia; Acute Lymphoblastic Lymphoma
Keywords: stem cell transplant; bone marrow transplant; transplantation conditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TBI: 200 Centigray (cGy) (Active Comparator): 200 cGy TBI is administered based on randomization in a single fraction on Day -3, -2, or -1, depending on if and how many days of rest are permitted.
  A day of rest occurring after preparative regimen completion and prior to stem cell infusion, is not routinely scheduled. Up to two days of rest may be added in this window based on logistical considerations or clinically as indicated. For one day of rest, TBI would be administered on Day -2. For two days of rest, TBI would be administered on Day -3.
  Interventions: Radiation: 200 cGy or 400 cGy total body irradiation (TBI)
- TBI: 400 cGy (Active Comparator): 400 cGy TBI is administered based on randomization in a single fraction on Day -3, -2, or -1, depending on if and how many days of rest are permitted.
  A day of rest occurring after preparative regimen completion and prior to stem cell infusion, is not routinely scheduled. Up to two days of rest may be added in this window based on logistical considerations or clinically as indicated. For one day of rest, TBI would be administered on Day -2. For two days of rest, TBI would be administered on Day -3.
  Interventions: Radiation: 200 cGy or 400 cGy total body irradiation (TBI)

INTERVENTIONS:
Radiation: 200 cGy or 400 cGy total body irradiation (TBI) — Either 200 or 400cGy will be given as part of reduced-intensity conditioning prior to consolidative allogeneic bone marrow transplant (alloBMT)

SUMMARY:
This is a randomized phase II trial of standard-of-care reduced-intensity conditioning (RIC) with 200 versus 400 cGy of total body irradiation (TBI) in patients with acute leukemia undergoing first allogeneic blood or marrow Transplantation (BMT). The primary objective is to compare the rates of graft-versus-host disease-free and relapse-free survival (GRFS) between patients in the two cohorts.

DETAILED DESCRIPTION:
This research is being done to learn more about reduced-intensity conditioning stem cell transplant for patients with acute leukemias or acute lymphoblastic lymphoma, using stem cell donation from the peripheral blood or bone marrow from a relative or an unrelated donor.

The purpose of this study is to determine if a TBI dose of 400 cGy yields better transplant-related outcomes than a TBI dose of 200 cGy when leukemia patients in remission undergo a reduced-intensity conditioning transplant using high-dose post-transplantation cyclophosphamide as GVHD prophylaxis. The study will use graft-versus-host disease-free, relapse-free survival (GRFS) as its primary endpoint. GRFS will be defined as time from transplant to the first of any grade III-IV acute GVHD, chronic GVHD requiring systemic immune suppression, disease relapse or progression, or death by any cause.

The transplantation of stem cells from the peripheral blood or bone marrow of a related or unrelated donor is a standard, established treatment for both acute leukemias and acute lymphoblastic lymphoma. Possible donors include parents, siblings, and children. The donor may also be unrelated to the patient. In order to help the donor cells grow, standard of care chemotherapy and radiation will be given before the transplant. Standard of care prophylactic immunosuppression will be used and includes the use of post-transplant cyclophosphamide. These medications lower the risk of GVHD and graft rejection. The exact planned duration of prophylactic immunosuppression will be dictated by institutional protocols based on donor type.

Reduced-intensity transplants have been given to many people in the treatment of various cancers. Over 1000 people at Johns Hopkins have received this type of transplant. Standard chemotherapy, commonly fludarabine and cyclophosphamide, along with radiation will be administered before infusion of the cells transplanted from the donor. The radiation administered as part of this pre-transplant conditioning regimen is called total body irradiation (TBI). This is important in allowing the donated stem cells to grow. TBI may also kill residual cancer cells. The optimal dose of TBI is unknown. Very high doses of TBI have been used previously and are associated with some anti-cancer activity but also significant side effects and an increased risk of death. Due to the significant risks associated with high doses of TBI, the practice at Johns Hopkins has been to use lower doses of TBI, either 200 or 400 centiGray (cGy) in one administration. It is unclear which of these doses, 200 or 400 centiGray (cGy), is superior in balancing anti-cancer effects and reducing side effects. The higher dose of TBI may increase the anti-cancer activity and the chance of engraftment, thereby reducing the patient's risk of disease relapse, which can be fatal. The lower dose of TBI may decrease the risk of blood transfusions, infertility, infections, GVHD, second cancers, and death without disease relapse.

The main goal of the study is to see which of these doses of TBI, 200 or 400 cGy, as part of reduced-intensity conditioning before stem cell transplantation, is superior in terms of reducing the combined risk of leukemia relapse, death, and severe GVHD. The study also looks at whether there is a difference in whether the donated stem cells engraft, time to blood count recovery, time admitted to a hospital, new cancers developing after stem cell transplant, overall severe side effects, how many people survive without cancer, and how many people survive overall depending on the dose of radiation received.

Patients will be randomly assigned to receive either 200 or 400 cGy of total body irradiation (TBI) as part of the reduced intensity conditioning regimen before stem cell transplant. This decision will be based a computer system that randomizes people into each group.

The study regimen includes several days of chemotherapy, immunosuppressant, and a single dose of radiation, either 200 or 400 cGy, followed by the bone marrow transplant. After the transplant, patients will receive two doses of the intravenous chemotherapy cyclophosphamide and two oral medications to prevent graft versus host disease and to aid in bone marrow engraftment. Participation on this study will last up to 2 years after transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 0 years
2. Patients with a diagnosis of acute myeloid leukemia (AML), acute lymphoblastic leukemia or lymphoma (ALL), or acute leukemia of mixed or ambiguous lineage per the 2022 World Health Organization classifications,75,76 with < 5% blasts on bone marrow morphologic analysis performed within 30 days of planned conditioning initiation

   1. AML is generally defined as ≥ 20% myeloid blasts identified in the peripheral blood and/or bone marrow. Myeloid sarcoma is also recognized as an AML-defining entity. Situations in which AML can be diagnosed without a specific blast threshold met nor myeloid sarcoma present are when fusions involving RUNX1::RUNX1T1, CBFB::MYH11, DEK:NUP214, or RBM15::MRTFA are present; rearrangements involving KMT2A, MECOM, or NUP98 exist; or there is a mutation in NPM1.
   2. B- or T-ALL is defined as the presence of lymphoid blasts identified in the peripheral blood and/or bone marrow with no specific blast threshold needed (acute lymphoblastic leukemia) or the presence of a lymphatic-based collection of lymphoblasts (acute lymphoblastic lymphoma).
   3. Acute leukemia of mixed or ambiguous lineage is defined as mixed or ambiguous lineage blasts identified in the peripheral blood and/or bone marrow or the presence of a lymphatic-based collection (lymphoma) of mixed or ambiguous lineage blasts. A specific blast threshold does not need to be met.
   4. Patients with a documented diagnosis of myeloproliferative neoplasm (MPN), myelodysplastic syndrome or neoplasm (MDS), and/or MDS/MPN-overlap prior to diagnosis of acute leukemia may be included for randomization in this clinical trial so long as the patient has received at least 4 cycles of DNA methyltransferase inhibitor (e.g., azacitidine, decitabine, decitabine/cedazuradine (Inqovi), and/or any other agent that works via this mechanism) or at least one cycle of induction chemotherapy. A list of antecedent diagnoses per the World Health Organization 2022 classification of hematolymphoid tumors that pertain to this inclusion criterion are listed below 75

      * i. MPN includes myelofibrosis, essential thrombocythemia, polycythemia vera, chronic neutrophilic leukemia, chronic eosinophilic leukemia, juvenile myelomonocytic leukemia, chronic myeloid leukemia (CML), or myeloproliferative neoplasm, not otherwise specified
      * ii. Myelodysplastic syndrome or neoplasm (MDS)
      * iii. MDS/MPN-overlap includes chronic myelomonocytic leukemia (CMML), myelodysplastic/myeloproliferative neoplasm with neutrophilia, myelodysplastic/myeloproliferative neoplasm with SF3B1 mutation and thrombocytosis, or myelodysplastic/myeloproliferative neoplasm, not otherwise specified
      * iv. Of note, patients without a documented history of one of these conditions prior to diagnosis of acute myeloid leukemia with myelodysplastic features would not be restricted to this specific criterion for study inclusion.
3. No active extramedullary leukemia or known active Central Nervous System (CNS) involvement by malignancy. Such disease treated into remission is permitted.
4. Patients must have a related or unrelated bone marrow or peripheral blood donor

   1. Human leukocyte antigen (HLA)-matched (10/10) sibling donor (MSD)
   2. HLA-matched (10/10) unrelated donor (MUD)
   3. HLA-haploidentical (5/10) related donor (Haplo)
   4. HLA-mismatched (6-9/10) unrelated donor (mMUD)
5. Planned allogeneic BMT using post-transplantation cyclophosphamide (PTCy) as a component of GVHD prophylaxis
6. Adequate end-organ function as measured by:

   1. Left ventricular ejection fraction greater than or equal to 35% or shortening fraction > 25%
   2. Bilirubin ≤ 3.0 mg/dL (unless due to Gilbert's syndrome or hemolysis), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 x Upper Limit of Normal (ULN)
   3. Forced Expiratory Volume in one second (FEV1) and Forced Vital Capacity (FVC) > 40% of predicted
7. Patients may enroll in other transplant-related trials (e.g., those testing post-transplant maintenance strategies or peri-transplant strategies for the management of donor specific antibodies) as long as other eligibility criteria are met and the requirements do not conflict with the treatment plan as outlined herein. Patients may also receive standard of care post-transplant maintenance therapies.

Exclusion Criteria:

1. Acute leukemia with promyelocytic leukemia (PML)/retinoic acid receptor α (RARA) fusion
2. Prior allogeneic BMT
3. Eastern Cooperative Oncology Group (ECOG) Performance Status > 2 or Karnofsky/Lansky score < 60
4. Patients with an additional active malignancy with a life expectancy < 2 years due to that disease
5. Symptomatic coronary artery disease
6. Uncontrolled infection
7. Patients who are pregnant or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
graft-versus-host disease-free, relapse-free survival (GRFS) | 2 years
  Number of patients without grade III-IV acute GVHD, chronic GVHD requiring systemic immune suppression, disease relapse or progression, or death by any cause from time of transplant until end of study

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  Number of patients surviving from day of transplant until end of study
Relapse-free survival (RFS) | 2 years
  Number of patients who are disease relapse free from time of transplant until end of study
Relapse Incidence | 2 years
  Cumulative incidence of relapse in each treatment arm from time of transplant until end of study
Non-relapsed mortality (NRM) | 2 years
  Number of people who died without disease relapse in each treatment arm from time of transplant until end of study
Graft vs Host Disease (GVHD)- moderate-to-severe chronic GVHD | 2 years
  Number of incidences of moderate-to-severe chronic GVHD from time of transplant until end of study
Graft vs Host Disease (GVHD)- acute grade II-IV | 2 years
  Number of incidences of acute grade II -IV GVHD from time of transplant until end of study
Graft vs Host Disease (GVHD)- grade III-IV | 2 years
  Number of incidences of grade III-IV GVHD from time of transplant until end of study
Graft Failure | 2 years
  Incidence of graft failure from time of transplant until end of study

OTHER OUTCOMES:
Incidence of Toxicities Grade ≥3 NCI CTCAE | Day 0 until Day +56
  Number of grade ≥ 3 toxicities occurring Grade ≥ 3 toxicities occurring from time of transplant until day +56
Incidence of Noninfective (Hemorrhagic Cystitis), Grade ≥2 NCI CTCAE | Day 0 until Day +56
  Number of grade ≥ 2 noninfective cystitis events occurring from time of transplant until day +56
Maximal Grade of Fatigue | Day 0 until Day +56
  maximal grade of fatigue according to the NCI CTCAE grading system from time of transplant until Day +56
Incidence of new malignancies | 2 years
  All malignancies newly diagnosed after beginning the conditioning regimen until end of study
Neutrophil engraftment | Day 0 until Day +28
  Cumulative incidences of neutrophil engraftment at 28 days
Platelet engraftment | Day 0 until Day +60
  Cumulative incidences of platelet engraftment at 60 days
Red Blood Cell (RBC) engraftment | Day 0 until Day +56
  The number of packed red blood cell (pRBC) transfusions administered
Degree of Donor Engraftment | 2 years
  median percentage of donor chimerism in total leukocytes and T cells at days 28, 56, 90, 180, 365, and 730
Comparison of scores between arms in Patient-Reported Health Outcomes Composite score | 2 years
  Scoring determined per the Research and Development (RAND) Corporation 36-Item Health Survey 1.0 (SF-36). The total score range from 0 to 100, with a higher score indicating better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Webster, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No